CLINICAL TRIAL: NCT00910234
Title: Early Treatment With Recombinant Erythropoietin for Neuroprotection in Very Preterm Infants: Comparison of High and Low Dose
Brief Title: Recombinant Erythropoietin for Neuroprotection in Very Preterm Infants
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Bai-Horng Su, MD, PhD., Chairman of Department of Pediatrics, China Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DMR-98
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Infant, Premature; Leukomalacia, Periventricular; Intraventricular Hemorrhage; Retinopathy of Prematurity
Keywords: Periventricular leukomalacia (PVL); Erythropoietin (EPO); Retinopathy of prematurity (ROP); Hypoxia-ischemia
MeSH Terms: conditions — Premature Birth; Leukomalacia, Periventricular; Retinopathy of Prematurity | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Drug: rhEpo, low dose (Active Comparator): rhEpo is administered 100 U/kg, iv at 3 to 6 hours after birth, and at 24 hours interval for another 2 doses.
  Interventions: Drug: recombinant human erythropoietin (rhEpo)
- Drug: rhEpo, high dose (Active Comparator): rhEpo is administered 3000 U/kg, iv at 3 to 6 hours after birth, and at 24 hours interval for another 2 doses.
  Interventions: Drug: recombinant human erythropoietin (rhEpo)
- Control Normal saline (Placebo Comparator): normal saline is administered 0.5/kg, iv at 3 to 6 hours after birth, and at 24 hours interval for another 2 doses.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: recombinant human erythropoietin (rhEpo) — rhEpo is administered 3000 U/kg, iv at 3 to 6 hours after birth, and at 24 hours interval for another 2 doses.
  Other Names: Epoietin Beta
  Arms: Drug: rhEpo, high dose
Drug: recombinant human erythropoietin (rhEpo) — rhEpo is administered 100 U/kg, iv at 3 to 6 hours after birth, and at 24 hours interval for another 2 doses.
  Other Names: Epoietin Beta
  Arms: Drug: rhEpo, low dose
Drug: Normal saline — normal saline is administered 0.5/kg, iv at 3 to 6 hours after birth, and at 24 hours interval for another 2 doses.
  Other Names: N/S solution
  Arms: Control Normal saline

SUMMARY:
Periventricular leukomalacia (PVL) is one of the most common brain injuries that occur in preterm infants. Inflammation, hypoxia-ischemia, free oxygen radical formation and excitotoxicity are all known pathogenic mechanisms that mediate this injury. Erythropoietin (EPO) has been shown to be protective against hypoxic-ischemic and inflammatory injuries. During the past decade, recombinant human Epo (rhEpo) has been widely used in preterm infants to prevent or treat the anemia of prematurity, in general, rhEpo has been considered to be safe and well tolerated in preterm infants. EPO was considered not capable of passing through blood-brain-barrier at low dose. Evidence from animal experiments reveals that rhEpo must be given in high doses at the beginning or within a short (up to 6 hours), critical time period after the onset of brain injury to achieve a significant neuroprotective effect. A recent study using high-dose rhEpo (3000 U rhEpo/kg body weight at birth) for neuroprotection in very preterm infants revealed that no signs of adverse effects of early high-dose rhEpo treatment in very preterm infants were identified. Contrary to this, a recent study in PVL of a rat model revealed that using a low dose rhEpo (50-100 U/kg) was effective in the treatment of brain damage induced by hypoxia-ischemia and did not affect normal oligodendrocyte maturity. On this basis, the researchers intent to investigate (1) whether low-dose rhEpo (100 U/kg) or high-dose rhEpo (3,000 U/kg) given to very preterm infants (gestation age < 32 weeks) immediately after birth and subsequently during the first 2 days is safe and possesses neuroprotective properties;(2) whether there are gender differences in response to the hypoxia-ischemic insult and EPO treatment; (3)the pharmacokinetics of low dose and high dose rhEPO. Very preterm infants with gestational age of < 32 weeks and admitted to the NICU are eligible for enrollment.

DETAILED DESCRIPTION:
Periventricular leukomalacia (PVL) is one of the most common brain injuries that occur in preterm infants. Inflammation, hypoxia-ischemia, free oxygen radical formation and excitotoxicity are all known pathogenic mechanisms that mediate this injury. Although several treatment strategies have been devised, few therapies effectively mitigate the harmful effects of hypoxia-ischemia in preterm newborns and the ensuing neurodevelopment sequelae. Erythropoietin (EPO) has been shown to be protective against hypoxic-ischemic and inflammatory injuries in neuronal cell culture, animal models of brain injury, and clinical trials of adult humans. During the past decade, recombinant human Epo (rhEpo) has been widely used in preterm infants to prevent or treat the anemia of prematurity, in general, rhEpo has been considered to be safe and well tolerated in preterm infants. EPO was considered not capable of passing through blood-brain-barrier at low dose. Evidence from animal experiments reveals that rhEpo must be given in high doses at the beginning or within a short (up to 6 hours), critical time period after the onset of brain injury to achieve a significant neuroprotective effect. A recent study using high-dose rhEpo (3000 U rhEpo/kg body weight at birth) for neuroprotection in very preterm infants revealed that no signs of adverse effects of early high-dose rhEpo treatment in very preterm infants were identified. Contrary to this, a recent study in PVL of a rat model revealed that using a low dose rhEpo (50-100 U/kg) was effective in the treatment of brain damage induced by hypoxia-ischemia and did not affect normal oligodendrocyte maturity. Clinical studies suggest that gender influences the response to brain injury. Ment and coworkers have reported that the cyclooxygenase inhibitor indomethacin ameliorated intraventricular hemorrhage and improved cognition in very low birth weight boys, but not girls. On this basis, the researchers intent to investigate (i) whether low-dose rhEpo (100 U/kg) or high-dose rhEpo (3,000 U/kg) given to very preterm infants (gestation age < 32 weeks) immediately after birth and subsequently during the first 2 days is safe and possesses neuroprotective properties; (ii) whether there are gender differences in response to the hypoxia-ischemic insult and EPO treatment; (iii)the pharmacokinetics of low dose and high dose rhEPO. Very preterm infants with gestational age of < 32 weeks and admit to our NICU are eligible for enrollment. After informed consent is obtained, infants will be randomly assigned to three groups based on a double-blind design. The study medication (rhEpo or NaCl 0.9%) is dispensed to each patient number that is blinded to the clinical investigators. Epoietin Beta or an equivalent volume of normal saline placebo is given intravenously during a period of 10 minutes at 3 to 6 hours after birth, and at 24 hours interval for another 2 doses.The primary short-term outcome measures are brain injury (intraventricular hemorrhage (IVH) and periventricular leukomalacia (PVL)) and ROP. The secondary outcomes are sepsis, necrotizing enterocolitis (NEC), persistent ductus arteriosus (PDA), apnea of prematurity, and chronic lung disease. The long term outcomes are whether early low-dose or high-dose treatment of rhEpo in very preterm infants finally improves neurodevelopmental outcome at 24 months' and 5 years' corrected age.

ELIGIBILITY:
Inclusion Criteria:

* After informed consent is obtained, very preterm infants with gestational age of < 32 weeks and admit to our NICU are eligible for enrollment.

Exclusion Criteria:

* Genetically defined syndromes,
* Congenital malformations that adversely affect neurodevelopment.

Ages: 2 Hours to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
The primary short-term outcome measures are brain injury (intraventricular hemorrhage (IVH) and periventricular leukomalacia (PVL)) and ROP. | 2 months

SECONDARY OUTCOMES:
The secondary outcomes are sepsis, necrotizing enterocolitis (NEC), persistent ductus arteriosus (PDA), apnea of prematurity, and chronic lung disease. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Bai-Horng Su, MD, PhD, Study Chair — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan